CLINICAL TRIAL: NCT01601444
Title: Detection of Pleural Effusion by Internal Thoracic Impedance Method
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Michal Roll PhD,MBA (Other Government)
Responsible Party: Sponsor-Investigator, Michal Roll PhD,MBA, Director, Research and Development, Tel-Aviv Sourasky Medical Center
Organization: Tel-Aviv Sourasky Medical Center (Other Government)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: TASMC-11-CG-504-CTIL
Record Dates: First submitted 2012-04-30; First posted 2012-05-18 (Estimated); Last update posted 2012-05-18 (Estimated); Status verified 2012-05

CONDITIONS: Pleural Effusion
Keywords: To assess pleural effusion by measuring internal thoracic impedance
MeSH Terms: conditions — Pleural Effusion | interventions — Electromyography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Pletysmograph — Pletysmograph electrodes are applied to the thoracic wall
  Other Names: Edema Guard Monitor (EMG) model RS-207 (RS Medical Monitoring Ltd. Jerusalem, Israel

SUMMARY:
Early detection of pleural effusion (PLE) would improve the treatment. However, preclinical detection of pleural effusion is often not possible.

Radiographic examination, widely used for detecting pleural effusion ,is not suitable for prolonged monitoring of patients at high risk of developing PLE especially ambulatory or at home The currently available methods for monitoring and early detection such as the measurement of pulmonary capillary wedge pressure or measurement by double indicator thermodilution, are not reliable enough and may themselves lead to complications.

Measuring internal thoracic impedance (ITI), the main component of which is lung impedance, is a noninvasive and safe method. PLE will be diagnosed in accordance with well-accepted clinical signs(dyspnea, cyanosis, pulmonary rales, crepitations, arterial hypoxemia) and roentgenological criteria

DETAILED DESCRIPTION:
Early detection of pleural effusion (PLE) would improve the treatment. However, preclinical detection of pleural effusion is often not possible.

Radiographic examination, widely used for detecting pleural effusion ,is not suitable for prolonged monitoring of patients at high risk of developing PLE especially ambulatory or at home (1-9).

The currently available methods for monitoring and early detection such as the measurement of pulmonary capillary wedge pressure or measurement by double indicator thermodilution, are not reliable enough and may themselves lead to complications(2-8).

Yu C-M et al.(9) recently reported successful prediction of CPE by a surgically implanted impedance plethysmograph integrated into a pacemaker . The system was shown to be sufficiently sensitive for cardiogenic pulmonary edema preceding. However this method is invasive and not suitable for wide use (9).

Therefore, these methods are seldom employed for the detection of PLE (3-7). Thus, a safe and accurate technique for early detection and monitoring of PlEf would be of great clinical value. The changes in the blood and extravascular fluid content in the lungs in humans and animals can be easily monitored using a noninvasive and totally safe procedure based on impedance plethysmography (5-12-). This method is based on the fact that the impedance of the lungs decreases with the increase in the fluid and free ions content in them (8,13,). However, it proved to be unsuitable for preclinical stage monitoring of PLE (2-8) for several reasons, mainly the low sensitivity of the existing impedance plethysmographs. This is due to the high skin-electrode contact resistance (13,14), which is of an order of magnitude high erthan the impedance of the lung.

After cleaning the skin of fats with alcohol and moistening it with electrode paste, the value of the skin electrode contact resistance is approximately 400- 500 ohm (11-13). Therefore, for two measuring electrodes (front and back of the chest), this value must be 800-1000 ohm.

Total transthoracic impedance (TTI) consists of internal thoracic impedance (ITI) and skin contact impedance. The TTI may vary from 920 to 1230 ohm in different individuals (11-13). However, change of TTI in PLE was reported by others to vary in the range of 2-16 ohm (7-9, 11-18), which is approximately1% of TTI and 1.5% of skin contact impedance. Monitors used in previous works were not sensitive enough to detect the relatively small changes in pulmonary impedance(2-7).

In addition, during prolonged monitoring, the skin-electrode contact impedance may also change (13,14) due to penetration of the ions from sweat into the electrode paste and drying of the paste. It may significantly exceed the change in the impedance of the lung caused by the development of cardiogenic pulmonary edema (2-7). Kubicek et al. (10) attempted to develop a method in which a tetrapolar electrode system is used to overcome this problem.

However, because this system measures the impedance of the entire chest, a large part of the electrical field is concentrated in the surface tissues, and this considerably reduces the sensitivity of the method (10,11). Furthermore, Kubicek's electrodes may be burdensome and for critically ill patients when prolonged monitoring is required. The main disadvantage of this and other more sensitive methods is surgical implantation of the electrodes (10,13) A new impedance monitor, model RS- 207 EDEMA GUARD MONITOR (R. S. Medical Monitoring, Jerusalem, Israel), has been developed (15). The monitor design has also solved the problem of the drift skin-to-electrode electrical resistance and its drift during prolonged monitoring by separating ITI from skin-to-electrode electrical resistance. The result of the above mentioned actions is a value of Internal Thoracic Electrical Resistance (Impedance) - ITI. The method of ITI estimation that completely described by Rabinovich (15) Unlike the existing impedance monitors, the new monitor measures only ITI, which roughly equals lung impedance, by automatically calculating skin electrode impedance and subtracting it from TTI. According to the published data, ITI ranges from 40 to 100 ohm in individuals without CPE and, on average, decreases to 30 ohm, i.e., by30% to 75% during CPE (11-12,16-21). These results showed much higher sensitivity compared with the 1.5% changes found using TTI methods. This is an average 35- fold increase (range, 20- to 50-fold intraindividual constitutional differences) of impedance plethysmograph sensitivity compared with the method without substraction of skin electrode resistance (2-8). This monitor was succefully used for early detection of pulmonary edema however there was no any expearence on pleural fluid detection.(11,12,16-20.) The aim of the present study is to evaluate the suitability of the RS-207 in monitoring PlEf at clinical and preclinical stage. The tests will be considered successful if ITI will be low or decreased parallel to or before the appearance of clinical signs and radiograph findings compatible with PlEf, and then demonstrably increased during their resolution.

Considerations and purpose Previous study based on measurements of ITI in early diagnosis of pulmonary edema showed suitability of the RS-207.

There is no any study that deals with early diagnosis of pleural effusion by this simple nonexpencive method which can be used in ICU and ambulatory Measuring ITI, the main component of which is lung impedance, is a noninvasive and safe method. PLE will be diagnosed in accordance with well-accepted clinical signs(dyspnea, cyanosis, pulmonary rales, crepitations, arterial hypoxemia) and roentgenological criteria.

The consideration of the study : evaluation of the suitability of the RS-205 monitor in detecting the PLE at preclinical stage before the appearance of clinical signs for assessment of early treatment and then to demonstrate increased of ITI during their resolution.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria for study group will be as follows: patients 40-90 year old with pleural effusion on chest X-ray of different etiologies:

  * coronary heart disease-(CHD)
  * valvular heart disease
  * renal failure
  * infectious disease malignant diseases( all complicated by pleural effusion).
* The control group will be comprised of patients 40-90years old without pleural effusion established by chest X-ray.

Exclusion Criteria:

* The exclusion criteria will be respiratory failure due to diseases, wearing a pacemaker,thoracic deformation, pulmonary edema and embolism

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2012-06; Primary Completion 2013-05 (Estimated); Study Completion 2013-08 (Estimated)

PRIMARY OUTCOMES:
Internal thoracic impedance | 12 months

REFERENCES:
- [Derived] Charach G, Rubalsky O, Charach L, Rabinovich A, Argov O, Rogowski O, George J. Internal thoracic impedance - a useful method for expedient detection and convenient monitoring of pleural effusion. PLoS One. 2015 Apr 28;10(4):e0122576. doi: 10.1371/journal.pone.0122576. eCollection 2014. PMID 25919389